CLINICAL TRIAL: NCT06117319
Title: Development and Validation of Sports Facilities in a Supportive Environment to Improve the Well-being of the Elderly
Brief Title: Immersive Technology and Virtual Reality as a Health Support Tool in a Residence for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); SEC Fonds Immobilier Groupe Maurice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RD-277_VR and elderly
Record Dates: First submitted 2023-09-13; First posted 2023-11-07 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Aging Well
Keywords: Aging well; virtual reality; activity; learning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 2 groups with different learning modalities (individual feedback compared to collective feedback)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual assistance (Experimental): 5 sessions with individual assistance
  The Virtual Reality (VR) activity will take the form of five (5) weekly training sessions.
  * Session 1(day 1): Basics of VR.
  * Session 2(day 8): 1-multiplayer game mode.
  * Session 3(day 15): Playing with a library. Browsing a library
  * Session 4(day 22): 2-individual game mode.
  * Session 5(day 29): Game practice.
  For each session, in small groups of 3 people, it will be proposed to test games requiring only movements of the upper limbs of low to moderate intensity. Sitting will be mandatory for the tests in order to avoid falls.
  Interventions: Other: Individual assistance Virtual reality training sessions
- Collective assistance (Experimental): 4 sessions with collective assistance and 1 session with individual assistance (session 5)
  The Virtual Reality (VR) activity will take the form of five (5) training sessions.
  * Session 1(day 1): Basics of VR.
  * Session 2(day 8): 1-multiplayer game mode.
  * Session 3(day 15): Playing with a library. Browsing a library
  * Session 4(day 22): 2-individual game mode.
  * Session 5(day 29): Game practice.
  For each session, in small groups of 3 people, it will be proposed to test games requiring only movements of the upper limbs of low to moderate intensity. Sitting will be mandatory for the tests in order to avoid falls.
  The collective assistance group was abandonned because tests revealed issues with ability of participants to help each other during VR sessions. No participants were ever assigned to this group.
  Interventions: Other: Collective assistance Virtual reality training sessions

INTERVENTIONS:
Other: Individual assistance Virtual reality training sessions — 5 virtual reality training sessions where feedback will be provided to each individual by the research team
  Arms: Individual assistance
Other: Collective assistance Virtual reality training sessions — 4 virtual reality training sessions where feedback will be provided to the whole group by the research team and 1 session where feedback will be individual. No participant was ever assigned to this intervention.
  Arms: Collective assistance

SUMMARY:
The purpose of this clinical trial is to learn more about the potential for using virtual reality in older adults living in residences for elderly to maintain health (physical activity, cognitive activity, social behaviors). The main questions it aims to answer are:

* To what extent can virtual reality be a tool to support health in older adults?
* What are the support needs of older adults in learning to use this immersive technology?

Participants are invited to complete 5 weekly training sessions on the use of a virtual reality headset. At the beginning and end of each session, participants will complete a questionnaire on their perception of their experience. During the sessions, the participants are asked to test games that mobilize the upper limbs. Two learning modalities are set up in two separate groups. These modalities aim to test two different support formulas in order to compare the support needs of the elderly in the use and integration of virtual reality to support the activities and health of this population.

ELIGIBILITY:
Inclusion Criteria:

* Independent person living in the sponsor's retirement home

Exclusion Criteria:

* Having a pacemaker
* Being at risk for epilepsy

Min Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Edith Martin, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participant was ever assigned to the collective assistance group.
Pre-assignment Details: The collective assistance group was abandonned because tests revealed issues with ability of participants to help each other during VR sessions.
Groups:
- Individual Assistance: 5 sessions with individual assistance
  The Virtual Reality (VR) activity will take the form of five (5) training sessions.
  * Session 1: Basics of VR.
  * Session 2: 1-multiplayer game mode.
  * Session 3: Playing with a library. Browsing a library
  * Session 4: 2-individual game mode.
  * Session 5: Game practice.
  For each session, in small groups of 3 people, it will be proposed to test games requiring only movements of the upper limbs of low to moderate intensity. Sitting will be mandatory for the tests in order to avoid falls.
  Individual assistance Virtual reality training sessions: 5 virtual reality training sessions where feedback will be provided to each individual by the research team
- Collective Assistance: The collective assistance group was abandonned because tests revealed issues with ability of participants to help each other during VR sessions. No participants were ever assigned to this group.
Period: Overall Study
Arm/Group | Individual Assistance | Collective Assistance
Started | 34 | 0
Completed | 34 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The collective assistance group was abandonned because tests revealed issues with ability of participants to help each other during VR sessions. No participants were ever assigned to this group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Assistance | Collective Assistance | Total
Number analyzed (Participants) | 34 | 0 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 34 |  | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 |  | 24
  Male | 10 |  | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 34 |  | 34
Region of Enrollment [Number; unit: participants]
  Canada | 34 |  | 34

OUTCOME MEASURES:

1. Primary Outcome: Learning of Virtual Reality Tasks
Description: Total score on 43 different tasks using a 5 point scale for each task(impossible(0), completion with external help(1), delay before individual completion and multiple repetitions(2), individual completion with less than 2 repetitions(3), individual completion without repetition(4) scored from 0 to 4 respectively). Scores for each session are averaged (Total score range from 0 to 4). Interpretations should be taken with caution(see Analysis population description).
Time Frame: During each 45 minutes intervention session on Session 1(Day 1), Session 2(Day 8), Session 3(Day 15), Session 4(Day 22), Session 5(Day 29)
Population: The evaluators were also tasked to provide assistance to the participants, if needed, during sessions. However, the amount of assistance needed by the participants was much higher than anticipated and hindered data collection. Each task and each participant were missing data. Some participants were missing data for up to 80% of all tasks for a session. As an example, for a particular task, only 7 participants provided data in session 1, whereas in session 3, 26 participants provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
score on a scale
  Session 1 | 2.13 (0.10) |
  Session 2: number analyzed (Participants) | 32 | 0
  Session 2 | 2.17 (0.08) |
  Session 3: number analyzed (Participants) | 28 | 0
  Session 3 | 2.22 (0.10) |
  Session 4: number analyzed (Participants) | 31 | 0
  Session 4 | 2.22 (0.15) |
  Session 5: number analyzed (Participants) | 28 | 0
  Session 5 | 2.28 (0.10) |

2. Primary Outcome: Ease
Description: Measurement of the perception of ease using a one item 5 point scale (higher score means higher ease during the session).Total score range from 1 to 5.
Time Frame: Immediately after each 45 minutes intervention session on Session 1(Day 1), Session 2(Day 8), Session 3(Day 15), Session 4(Day 22), Session 5(Day 29)
Population: Number of participants analyzed for each session varies based on the number of participants present that day. Since group session were scheduled, absent participants couldn't complete the session later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
units on a scale
  Session 1(day 1) | 4.06 (1.01) |
  Session 2(day 8): number analyzed (Participants) | 32 | 0
  Session 2(day 8) | 3.53 (1.16) |
  Session 3(day 15): number analyzed (Participants) | 28 | 0
  Session 3(day 15) | 4.11 (1.03) |
  Session 4(day 22): number analyzed (Participants) | 31 | 0
  Session 4(day 22) | 3.58 (1.18) |
  Session 5(day 29): number analyzed (Participants) | 28 | 0
  Session 5(day 29) | 4.00 (1.19) |

3. Primary Outcome: Sense of Control: Measurement of the Participants' Sense of Control Using a Scale From 1 to 5
Description: measurement of the perception of sense of control using a one item 1-5 point scale (higher score means higher sense of control during the session).Total score range from 1 to 5.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
units on a scale
  Session 1(day 1) | 3.85 (0.82) |
  Session 2(day 8): number analyzed (Participants) | 32 | 0
  Session 2(day 8) | 3.53 (0.92) |
  Session 3(day 15): number analyzed (Participants) | 28 | 0
  Session 3(day 15) | 3.57 (0.96) |
  Session 4(day 22): number analyzed (Participants) | 31 | 0
  Session 4(day 22) | 3.19 (1.14) |
  Session 5(day 29): number analyzed (Participants) | 28 | 0
  Session 5(day 29) | 3.79 (1.07) |

4. Primary Outcome: Satisfaction With Supervision
Description: measurement of the perception of satisfaction using a one item 5 point scale (higher score means higher satisfaction during the session). Total score range from 1 to 5.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
score on a scale
  Session 1(day 1) | 4.76 (0.61) |
  Session 2(day 8): number analyzed (Participants) | 32 | 0
  Session 2(day 8) | 4.41 (0.95) |
  Session 3(day 15): number analyzed (Participants) | 28 | 0
  Session 3(day 15) | 4.68 (0.26) |
  Session 4(day 22): number analyzed (Participants) | 31 | 0
  Session 4(day 22) | 4.35 (0.95) |
  Session 5(day 29): number analyzed (Participants) | 29 | 0
  Session 5(day 29) | 4.93 (0.37) |

5. Secondary Outcome: Stress Level at the Start of the Session
Description: Measurement of the participants' stress level using a 1-item scale from 1 to 5 (lower score means higher stress), total scale range is 1 to 5
Time Frame: Immediately before each 45 minutes intervention session on Session 1(Day 1), Session 2(Day 8), Session 3(Day 15), Session 4(Day 22), Session 5(Day 29)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
score on a scale
  Session 1(day 1) | 4.38 (0.85) |
  Session 2(day 8): number analyzed (Participants) | 32 | 0
  Session 2(day 8) | 4.78 (0.55) |
  Session 3(day 15): number analyzed (Participants) | 28 | 0
  Session 3(day 15) | 4.89 (0.42) |
  Session 4(day 22): number analyzed (Participants) | 30 | 0
  Session 4(day 22) | 4.77 (0.50) |
  Session 5(day 29): number analyzed (Participants) | 29 | 0
  Session 5(day 29) | 4.76 (0.44) |

6. Secondary Outcome: Desire to Play Virtual Reality Games
Description: number of participants mentionning the desire to play virtual reality games
Time Frame: as for outcome 2
Population: The collective assistance group was abandonned because tests revealed issues with ability of participants to help each other during VR sessions. No participants were ever assigned to this group.
  Number of participants analyzed for each session varies based on the number of participants present that day. Since group session were scheduled, absent participants couldn't complete the session later.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Assistance | Collective Assistance
Number analyzed (Participants) | 34 | 0
Participants
  Session 1(Day 1) | 4 |
  Session 2(Day 8): number analyzed (Participants) | 32 | 0
  Session 2(Day 8) | 3 |
  Session 3(Day 15): number analyzed (Participants) | 28 | 0
  Session 3(Day 15) | 2 |
  Session 4(Day 22): number analyzed (Participants) | 31 | 0
  Session 4(Day 22) | 4 |
  Session 5(Day 29): number analyzed (Participants) | 30 | 0
  Session 5(Day 29) | 9 |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the protocol wich took 29 days.
Description: No participants were ever assigned to the collective assistance group.
Arm/Group | Individual Assistance | Collective Assistance
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/0
Other Adverse Events (participants affected / at risk) | 0/34 | 0/0

LIMITATIONS AND CAVEATS:
The collective assistance group was abandoned because tests revealed issues with the ability of participants to help each other during VR sessions. No participants were ever assigned to this group.

Primary outcome 1 has a 80% missing data ratio for some tasks, futhermore missing data was present in all participants. Interpretations should be taken with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT06117319/Prot_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT06117319/ICF_001.pdf